CLINICAL TRIAL: NCT02352987
Title: Randomized, Single Blind, Placebo Controlled Clinical Trial to See the Effect of Combination of Neem, Propylene Glycol and Salicylic Acid in the Treatment of Arsenical Palmar Keratosis
Brief Title: Effect of Neem Extract, Propylene Glycol and Salicylic Acid Combination in the Treatment of Arsenical Palmar Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Prof., Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSMMU-008-CT
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Arsenic Poisoning
MeSH Terms: interventions — Propylene Glycol; Salicylic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients treated with 3 drugs (Experimental): Neem plus propylene glycol plus salicylic acid: Neem extract, propylene glycol (40%) and salicylic acid (10%) once daily on palm for 12 weeks
  Interventions: Drug: Neem plus propylene glycol plus salicylic acid
- Patients treated with 1 drug (Active Comparator): Salicylic acid once daily on palm for 12 weeks
  Interventions: Drug: Salicylic acid

INTERVENTIONS:
Drug: Neem plus propylene glycol plus salicylic acid — Leaf extract of neem plus propylene glycol (40%) plus salicylic acid (10%) will be applied on palmar keratotic lesion once daily at bedtime for 12 weeks
  Other Names: In house prepared
  Arms: Patients treated with 3 drugs
Drug: Salicylic acid — salicylic acid (10%) will be applied on palmar keratotic lesion once daily at bedtime for 12 weeks
  Other Names: In house prepared
  Arms: Patients treated with 1 drug

SUMMARY:
This study is designed to find out the effectiveness of combination of ethanol extract of neem leaf, propylene glycol (40%) and salicylic acid (10%) in the treatment of palmar arsenical keratosis.

DETAILED DESCRIPTION:
Arsenic, a non-essential trace element, is a major water pollutant in Bangladesh. Arsenical keratosis, which occurs in the palm and sole, is a common symptom of arsenicosis. The objective of this study is to find the effectiveness of combination of topical administration of the ethanol extract of leaf of neem (Azadirachta indica), propylene glycol (40%) and salicylic acid (10%) in the treatment of palmar arsenical keratosis. On the basis of inclusion and exclusion criteria, 30 patients of moderate palmar arsenical keratosis will be recruited from an arsenic affected area. They will be divided into two groups: study group and placebo comparator group. Each group consisting of 15 members. Study group will be given combination of ethanol extract of leaf of neem, propylene glycol (40%) and salicylic acid (10%) to apply on palm overnight once daily for 12 weeks. On the other hand placebo comparator group will be given salicylic (10%) acid to apply on palm overnight once daily for 12 weeks. Water and nail samples will be collected before starting recruitment to confirm arsenicosis. After conclusive recruitment of the subjects the objective, nature, purpose and potential risks and benefits of all procedures of the study will be explained in details to the patients and informed written consent will be taken from them. Detail history, clinical examination and photograph (palm) will also be collected. Clinical improvement will be assessed by measuring palmar nodular size on both hands, before starting treatment and after 12 weeks completion of treatment and perception of patients about their improvement. The study will explore the effectiveness of topical use of combination of ethanol extract of neem, propylene glycol and salicylic acid for the treatment of palmar arsenical keratosis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* Palmar arsenical keratosis
* Drinking arsenic contaminated water (>50 µg/L) for more than six months
* Patient voluntarily agree to participate

Exclusion Criteria:

* Pregnancy and lactating mother
* Skin lesion :Psoriasis and eczema
* Bowen's disease
* Any kind of systemic disease, inflammatory disease and infectious condition that affect skin (Diabetes mellitus, Rheumatoid arthritis, Systemic lupus erythematosus , Hepatitis and Tuberculosis)
* Hypersensitivity to any drug
* Patient who received treatment within last three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in palmer arsenical keratosis | 0 weeks (baseline), 12 weeks (end)
  Size of keratotic lesion will be decreased

SECONDARY OUTCOMES:
Changes in arsenic level in nail | 0 weeks (baseline), 12 weeks (end)
  Arsenic level in nail will be decreased

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Muradnagar Health Complex, Comilla, Bangladesh